CLINICAL TRIAL: NCT01643408
Title: Phase II, An Open Label, Single Arm, Multi-Center Pharmacokinetic Study of Intravenous Erwinaze (Asparaginase Erwinia Chrysanthemi)Following Allergy to Native E. Coli Asparaginase (Elspar or Kidrolase), Pegaspargase (Oncaspar) or Calaspargase Pegol (EZN-2285) in Children, Adolescents and Young Adults With Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma.
Brief Title: A Study of Erwinaze Administered Intravenously in Patients Who Had an Allergy to Frontline Asparaginase Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100EUSA12
Record Dates: First submitted 2012-06-25; First posted 2012-07-18 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Erwinaze; asparaginase; Eusa Pharma; Pharmacokinetic study; NSAA
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Erwinaze (Experimental)
  Interventions: Drug: asparaginase Erwinia chrysanthemi

INTERVENTIONS:
Drug: asparaginase Erwinia chrysanthemi

SUMMARY:
This study will utilize Erwinaze via intravenous administration in patients between the ages of 1 and 30 who have experienced an allergy to their frontline therapy. The study will determine the proportion of patients with 2 day nadir serum asparaginase activity levels that are >0.1 IU/mL during the first 2 weeks of treatment with 3 times per week IV dosing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma,
* Ages >/= 1 and </= to 30 years at the time of initial diagnosis
* Undergoing asparaginase treatment for ALL or lymphoblastic lymphoma
* Documented Grade 2 or higher hypersensitivity reaction to native or pegylated E. coli asparaginase or Calaspargase pegol
* Must have two remaining weeks of native E. coli asparaginase treatment or 1 remaining dose of either Pegaspargase or Calaspargase pegol
* Direct bilirubin less than or equal to Grade 2
* Amylase and lipase within normal limits (per institutional standards)
* Signed informed consent by the patient is greater than or equal to 18 years or by the parent if the patient is younger than 18 years old.

Exclusion Criteria:

-

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Vrooman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (22):
- United States (18):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange County, California
  - Stanford Medical Center, Palo Alto, California
  - Children's Hospital, Aurora, Colorado
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - John Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - UMDNJ/Robert Wood Johnson, New Brunswick, New Jersey
  - Columbia Presbyterian Medical Center, New York, New York
  - Montifiore Medical Center, The Bronx, New York
  - Oregon Health & Sciences, Portland, Oregon
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Inova Fairfax Medical Center, Falls Church, Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - McMasters University Medical Center, Hamilton, Ontario
  - Sick Children's Hospital, Toronto, Ontario
  - Hospital St. Justine, Saint Catherine, Quebec
  - Quebec Children's Hospital, Sainte-Foy, Quebec

REFERENCES:
- [Derived] Vrooman LM, Kirov II, Dreyer ZE, Kelly M, Hijiya N, Brown P, Drachtman RA, Messinger YH, Ritchey AK, Hale GA, Maloney K, Lu Y, Plourde PV, Silverman LB. Activity and Toxicity of Intravenous Erwinia Asparaginase Following Allergy to E. coli-Derived Asparaginase in Children and Adolescents With Acute Lymphoblastic Leukemia. Pediatr Blood Cancer. 2016 Feb;63(2):228-33. doi: 10.1002/pbc.25757. Epub 2015 Sep 16. PMID 26376459

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Population: All participants who received at least 1 dose of Erwinaze
Period: Overall Study
Arm/Group | Safety Population
Started | 30
Completed | 16
Not Completed | 14
Not completed — Adverse Event | 12
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: All patients who received at least one dose of Erwinaze
Arm/Group | Safety Population
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (5.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Two Day Nadir Serum Asparaginase Activity (NSAA) Level
Description: To report the mean 2 day NSAA levels (48 hour levels taken after the 5th dose) that are > or = 0.1 IU/mL during the first 2 weeks of treatment with 3-times per week intravenous dosing of Erwinase at 25,000 IU/m2/dose.
Time Frame: 48 hours post-dose 5
Population: The Pharmacokinetic (PK) population consisted of all participants who received at least 1 dose of Erwinaze and were considered evaluable.
Measure: Mean (Standard Deviation); unit: (IU/mL)
Groups:
- Open-Label Erwinaze: asparaginase Erwinia chrysanthemi
Arm/Group | Open-Label Erwinaze
Number analyzed (Participants) | 24
(IU/mL) | 0.32 (0.23)

2. Secondary Outcome: Proportion of Participants Achieving Sustained NSAA Values of >0.1 U/mL at 48 Hours
Description: To report the proportion of participants achieving 2 day NSAA levels (48 hour levels taken after the 5th dose) that are > or = 0.1 IU/mL during the first 2 weeks of treatment with 3-times per week intravenous dosing of Erwinase at 25,000 IU/m2/dose.
Time Frame: 48 hours post-dose 5
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Erwinaze
Number analyzed (Participants) | 24
Participants | 20

3. Secondary Outcome: Three Day NSAA Level
Description: To report the mean 3 day NSAA levels (72 hour levels taken after the 6th dose) that are > or = 0.1 IU/mL in the first 2 weeks of treatment with 3 times per week intravenous dosing of Erwinase at 25,000 IU/m2/dose.
Time Frame: 72 hours post-dose 6
Measure: Mean (Standard Deviation); unit: (IU/mL)
Arm/Group | Open-Label Erwinaze
Number analyzed (Participants) | 21
(IU/mL) | 0.09 (0.07)

4. Secondary Outcome: Proportion of Participants Achieving Sustained NSAA Values of >0.1 U/mL at 72 Hours
Description: To report the proportion of participants achieving 3 day NSAA levels (72 hour levels taken after the 6th dose) that are > or = 0.1 IU/mL in the first 2 weeks of treatment with 3 times per week intravenous dosing of Erwinase at 25,000 IU/m2/dose.
Time Frame: 72 hours post-dose 6
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Erwinaze
Number analyzed (Participants) | 21
Participants | 9

5. Secondary Outcome: Nadir Serum Asparaginase Activity Over Time
Description: To describe the NSAA over time in participants with ALL/Lymphoblastic Lymphoma who have/had developed hypersensitivity to native E. coli asparaginase, Pegaspargase or Calaspargase pegol and are receiving intravenous Erwinaze 3 times per week for a prolonged duration (4-30 weeks).
Time Frame: 4 weeks to 30 weeks
Population: This population consisted of participants who completed Course 4 with Pharmacokinetic(s) (PK) assessments 48 hours after dose 5 (week 8).
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Open-Label Erwinaze
Number analyzed (Participants) | 6
IU/mL | 0.51 (0.252)

ADVERSE EVENTS:
Time Frame: 4 Weeks
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 15/30
Other Adverse Events (participants affected / at risk) | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=30)
Hypersensitivity (Immune system disorders) | 4
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 4
Pyrexia (General disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Bacteraemia (Infections and infestations) | 1
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Sepsis (Infections and infestations) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=30)
Hypersensitivity (Immune system disorders) | 10
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 4
Pyrexia (General disorders) | 3
Alanine Aminotransferase Increased (Investigations) | 3
Pancreatitis (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.